CLINICAL TRIAL: NCT00170196
Title: The CAPISCE-Trial: Community-Acquired Pneumonia; an Intervention Study With Corticosteroids
Brief Title: Efficacy Studies of Corticosteroid Therapy in Community-Acquired Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Center Alkmaar (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M05-018
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2008-09-29 (Estimated); Status verified 2008-09

CONDITIONS: Pneumonia
Keywords: pneumonia; corticosteroids
MeSH Terms: conditions — Pneumonia | interventions — Prednisone

INTERVENTIONS:
Drug: prednisone

SUMMARY:
The purpose of this study is to determine the efficacy of addition of corticosteroid therapy to antibiotics in patient admitted with Community-acquired pneumonia.

The hypothesis is: Prednisolone in combination with antibiotic treatments is effective in improving clinical outcome in patients hospitalized with CAP.

DETAILED DESCRIPTION:
Community-acquired pneumonia (CAP) is a acute illness with a considerable morbidity and mortality, especially patients with severe CAP. In the past decennia, in spite of many investigations, little reduction is seen in morbidity an mortality. Corticosteroids have a immune-modulation effect, which is not completely elucidated. Most likely the immune modulation effect is due to down-regulation of pro-inflammatory cytokines. The use of corticosteroids next to antibiotics in CAP could lead to shorter time to clinical stability, length of stay and costs.

Comparison: Hospitalized patients with CAP treated with antibiotics and prednisolone versus hospitalized patients with cap treated with antibiotics and placebo

ELIGIBILITY:
Inclusion Criteria:

Clinical symptoms of community-acquired pneumonia:

* Fever, cough, sputum, pleural pain, dyspnoea
* Radiological symptoms of pneumoniä

Exclusion Criteria:

* Any conditions wich requires corticosteroid therapy.
* Pregnancy of lactation
* Malignancy
* Immune-compromised patients (eg chemotherapy or AIDS)
* Pre-treatment with macrolide for >24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2005-08; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy at the end of treatment

SECONDARY OUTCOMES:
Clinical efficacy at follow up
Inflammation response (serummarkers)
Length of Stay
Time to clinical stability
Mortality
Time to defeverescence

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Snijders, Drs, Principal Investigator — Pulmo Science; Wim G Boersma, dr, Study Director — Pulmo Science
Locations (1):
- Medisch Centrum Alkmaar, Alkmaar, North Holland, Netherlands

REFERENCES:
- [Derived] Raeven VM, Spoorenberg SM, Boersma WG, van de Garde EM, Cannegieter SC, Voorn GP, Bos WJ, van Steenbergen JE; Alkmaar study group; Ovidius study group. Atypical aetiology in patients hospitalised with community-acquired pneumonia is associated with age, gender and season; a data-analysis on four Dutch cohorts. BMC Infect Dis. 2016 Jun 17;16:299. doi: 10.1186/s12879-016-1641-9. PMID 27317257
- [Derived] Snijders D, Daniels JM, de Graaff CS, van der Werf TS, Boersma WG. Efficacy of corticosteroids in community-acquired pneumonia: a randomized double-blinded clinical trial. Am J Respir Crit Care Med. 2010 May 1;181(9):975-82. doi: 10.1164/rccm.200905-0808OC. Epub 2010 Feb 4. PMID 20133929